CLINICAL TRIAL: NCT06190392
Title: Effect of a Global Simplified Strategy on Thromboembolic Events in Emergency Department Patients with Suspected Pulmonary Embolism
Acronym: MODS STRATEGY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP230886; 2023-A01956-39 (Other: IDRCB ANSM)
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Emergency department; PERC Rule
MeSH Terms: conditions — Pulmonary Embolism; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Modified simplified diagnostic strategy MODS (Experimental)
  Interventions: Other: MODS Modified simplified diagnostic strategy

INTERVENTIONS:
Other: MODS Modified simplified diagnostic strategy — The intervention will be the patient's management with a simplified global strategy. Whether PE is the most likely diagnostic will be assessed by the unstructured implicit clinician's estimation.
  In patient with a clinical suspicion of pulmonary embolism: DDimer testing will be performed.
  If the likelihood of PE is low (PE is not the most likely diagnosis), then threshold for DDimer testing will be 1000 ng/ml. If the likelihood of PE is high (PE is the most likely diagnosis), then the age-adjusted DDimer threshold will be applied.

SUMMARY:
Pulmonary embolism (PE) is frequently suspected in emergency departments (ED) patients which often leads to the prescription of DDimer testing and irradiative chest imaging (Computed Tomographic Pulmonary Angiogram CTPA in most cases).[1] Indeed, an increased use of CTPA has been reported without clear benefit in terms of prognosis.This increased use is reportedly associated with potential overdiagnosis of PE, increased cost, length of ED stay, and side effects from both chest imaging and undue anticoagulant treatments. The standard diagnostic strategy for PE work up includes three steps with an initial evaluation of clinical probability, followed by D-dimer testing if indicated, followed by chest imaging if necessary - Computed tomographic pulmonary angiogram CTPA being the imaging modality of choice.

A large European prospective study has reported that the use of CTPA has constantly increased without change in the diagnostic yield. In order to reduce the use of CTPA, it has been validated that in patients with a low likelihood of PE, the D-dimer threshold for ordering CTPA can be raised at 1000 ng/ml. It has been validated that a low likelihood of PE can be determined either with the YEARS or the PEGeD clinical decision rules. These latter two include one common item being "Is PE the most likely diagnosis". A retrospective cohort study of 3330 patients reported that using this sole question of "Is PE the most likely diagnosis" can be safely used to raise the D-dimer threshold to 1000 ng/ml, and that this performs as well as YEARS and PEGeD. This simple question is easier to use by emergency physicians compared to complex ones, which are reportedly seldom used by emergency physicians. Therefore, the validation of the "PE unlikely" simple and straightforward decision rule could increase physicians' adherence and therefore limit the use of chest imaging.

The hypothesis of this prospective study is that the likelihood of PE assessed to elevate the DDimer threshold to 1000 ng/ml can be estimated by the sole question of "is PE the most likely diagnosis", and to validate a global simplified diagnostic strategy for PE in the ED.

The intervention will be the patient's management with a simplified global strategy. Whether PE is the most likely diagnostic will be assessed by the unstructured implicit clinician's estimation.

In patient with a clinical suspicion of pulmonary embolism: DDimer testing will be performed.

If the likelihood of PE is low (PE is not the most likely diagnosis), then threshold for DDimer testing will be 1000 ng/ml. If the likelihood of PE is high (PE is the most likely diagnosis), then the age-adjusted DDimer threshold will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ED adult patients with suspected pulmonary embolism defined as:

  * New onset of or worsening shortness of breath
  * Or Chest pain
  * Or Syncope in the absence of any obvious other cause (such as pneumothorax, asthma attack, ST elevation myocardial infarction, trauma, etc.)
* Patient able to understand and give oral consent
* Informing and obtaining the patient's oral consent
* Social security affiliation (except AME)

Exclusion Criteria:

* Patients currently treated with full-dose anticoagulant therapy
* Diagnosed thrombo-embolic event in the past 6 months
* PE ruled out by the PERC rule (low clinical probability and none of the 8 items of the PERC score)
* Acute severe presentation (clinical signs of respiratory distress, hypotension, SpO2 < 90%, shock)
* DDimer level known before ED visit
* Patient living in assisted-living home or nursing home or palliative center. Anticipated life expectancy < 3 months or "do not resuscitate" order
* Patient under legal protection measure (tutorship or curatorship) and patient deprived of freedom
* Pregnancy and breastfeeding
* Participation in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1223 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
The failure proportion of the diagnostic strategy, defined as a diagnosed thrombo-embolic event at 3 months follow-up (either a PE or a deep venous thrombosis), among patients in whom PE was initially ruled out. | 3 months

SECONDARY OUTCOMES:
Pulmonary embolism | 3 months
Deep venous thrombosis | 3 months
CTPA or V/Q scan ordered by ED physicians | 3 months
Type of PE (lobar, segmental, sub-segmental) | 3 months
Hospital admission following the ED visit | 3 months
Anticoagulant therapy administration, | 3 months
All-cause mortality | 3 months
All-cause readmissions at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Héloïse BANNELIER, MD, MSc, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emergency department Hospital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Roussel M, Bannelier H, Lebal S, Kassasseya C, Bouzid D, Peyrony O, Baud A, Chauvin A, Beauvais A, Javaud N, Gorlicki J, Truchot J, Le Borgne P, Chocron R, Simon T, Freund Y. D-Dimer thresholds for diagnosis of pulmonary embolism based on a single question: is it the most likely diagnosis? A prospective, multicentre, open-label, single-arm interventional study. Lancet Respir Med. 2026 Jan;14(1):29-37. doi: 10.1016/S2213-2600(25)00292-9. Epub 2025 Oct 21. PMID 41135553